CLINICAL TRIAL: NCT04617730
Title: Randomized Trial to Quantify the Efficacy of the Safetac® Product Mepitel® Film on the Prevention of Radiodermatitis in the Inguinal Fold.
Brief Title: Efficacy of the Mepitel® Film on the Prevention of Radiodermatitis in the Inguinal Fold.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CE3220.
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Radiodermatitis; Radiation Toxicity; Radiotherapy Side Effect
Keywords: Radiodermatitis; Mepitel film; Inguinal fold; Radiotherapy
MeSH Terms: conditions — Radiodermatitis; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Active Comparator)
  Interventions: Other: Flamigel®
- Interventional arm (Experimental)
  Interventions: Device: Mepitel® film

INTERVENTIONS:
Device: Mepitel® film — This study is a comparative study between the standard procedure, which is to prescribe a hydro-active colloidal gel called Flamigel® to be applied to the irradiated area, and the use of Mepitel® Film.
  Arms: Interventional arm
Other: Flamigel® — The control arm will be treated according to the standard of care.
  Arms: Control arm

SUMMARY:
The aim is to quantify the efficiency of the Safetac product Mepitel® Film on the prevention of radiodermatitis for cancer patients treated with external beam radiation therapy near the inguinal fold(s). Previous studies have looked into the differences in skin reactions for Mepitel® Film versus hydro-active colloid gel in breast cancer [1, 2] and head and neck cancer [3]. In breast cancer, the prevalence of radiation induced dermatitis has strongly decreased due to of modern radiotherapy techniques and fractionation. In the groin, however, this is not the case, and radiation dermatitis remains an important problem. To the best of our knowledge, no previous study has looked into the efficiency of a prophylactic Mepitel® Film protocol in the inguinal fold. The goal of this study is to evaluate whether the Mepitel® Film offers a lower degree of radiation-induced dermatitis compared to hydro-active colloid gel and thereby challenging the gold standard.

References:

1. Herst, P., Bennett, N., Sutherland, A., Peszynski, R., Paterson, D. and Jasperse, M. (2014). Prophylactic use of Mepitel Film prevents radiation-induced moist desquamation in an intra-patient randomised controlled clinical trial of 78 breast cancer patients. Radiotherapy and Oncology, 110(1), pp.137-143.
2. Møller, P., Olling, K., Berg, M., Habæk, I., Haislund, B., Iversen, A., Ewertz, M., Lorenzen, E. and Brink, C. (2018). Breast cancer patients report reduced sensitivity and pain using a barrier film during radiotherapy - A Danish intra-patient randomized multicentre study. Technical Innovations & Patient Support in Radiation Oncology, 7, pp.20-25.
3. Wooding, H., Yan, J., Yuan, L., Chyou, T., Gao, S., Ward, I. and Herst, P. (2018). The effect of Mepitel Film on acute radiation-induced skin reactions in head and neck cancer patients: a feasibility study. The British Journal of Radiology, 91(1081), p.20170298.

ELIGIBILITY:
Inclusion Criteria:

* Patients with external beam radiotherapy of the bilateral inguinal nodal region, with at least 25 fractions of 1.8-2Gy per fraction.

Exclusion Criteria:

* Re-irradiation.
* Pregnancy.
* Patients under the age of 18.
* Patients not willing to participate (no informed consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevention of grade 2.5 RTOG radiodermatitis | Post 25 sessions
  To evaluate and quantify the influence of the Mepitel® Film dressing on the prevention of patchy moist desquamation (grade 2.5 RTOG) radiodermatitis in the inguinal fold.

SECONDARY OUTCOMES:
Time to radiodermatitis apparition | At the end of treatment
  To analyze the time it takes for the patchy moist desquamation (grade 2.5 RTOG) to appear and to evaluate whether it occurs later in the Mepitel® Film group.
Healing time | 3 months post treatment
  To analyze the time that the patchy moist desquamation takes to heal and to evaluate if the Mepitel® film group can heal faster.

IPD SHARING:
Plan to Share IPD: No